CLINICAL TRIAL: NCT00516412
Title: Master Protocol for Mantle Cell Lymphoma A Multicenter Phase II Trial Testing Everolimus (RAD001) for the Treatment of Patients With Relapsed or Therapy Resistant Mantle Cell Lymphoma
Brief Title: Everolimus in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 36/06; EU-20749; 2007-001108-19 (EudraCT Number)
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Genetic: molecular response by PCR

INTERVENTIONS:
Drug: everolimus — Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: RAD001
Genetic: molecular response by PCR — Bone marrow and peripheral blood samples are collected periodically and analyzed for molecular response by PCR. Molecular studies are also performed on DNA level formalin-fixed paraffin-embedded tissue

SUMMARY:
RATIONALE: Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluation of the efficacy and tolerability of everolimus in patients with relapsed or therapy-resistant mantle cell lymphoma.

Secondary

* Evaluation of the efficacy of everolimus to induce molecular remission in patients treated with this regimen.
* Investigation of immunoglobulin heavy chain variable gene somatic hypermutations (Ig-V_H) in classical mantle cell lymphoma as compared to blastoid mantle cell lymphoma, in particular in regard to their frequency, mutation distribution pattern (antigen selected vs. at random), and the individually involved Ig-V_H families.
* Evaluation of a putative impact of Ig-V_H on clinical outcome.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Bone marrow and peripheral blood samples are collected periodically and analyzed for molecular response by PCR. Molecular studies are also performed on DNA level formalin-fixed paraffin-embedded tissue samples.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed relapsed or chemotherapy/immunotherapy-resistant mantle cell lymphoma

  * No more than 3 lines of prior systemic treatment
* At least one measurable lesion ≥ 15 mm in its greatest transverse diameter by CT scan

Exclusion criteria:

* Presence or history of CNS disease (either CNS lymphoma or lymphomatous meningosis)
* Newly diagnosed mantle cell lymphoma
* Patients suitable for intensive treatment (e.g., hyperfractionated cyclophosphamide, vincristine, doxorubicin hydrochloride and dexamethasone with high-dose methotrexate and cytarabine [HyperCVAD])

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status ≤ 2
* Creatinine clearance ≥ 30mL/min
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* AST and ALT ≤ 2 times ULN
* Neutrophils ≥ 1,500/mm³ (≥ 1,000/mm³ with marrow infiltration)
* Thrombocytes ≥ 100,000/mm³ (≥ 75,000/mm³ in case of bone marrow infiltration)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after study participation

Exclusion criteria:

* Prior or concurrent hematological malignancies

  * Patients with prior solid organ tumors that required no treatment over the last 5 years and are currently free of disease are eligible
* Cardiovascular disease including any of the following:

  * NYHA class III or IV congestive heart failure
  * Unstable angina pectoris
  * Significant arrhythmia or arrhythmia requiring chronic treatment
  * Myocardial infarction in the last 3 months
* Serious underlying medical condition which could impair the ability of the patient to participate in the trial including any of the following:

  * Uncontrolled diabetes mellitus
  * Gastric ulcers
  * Active autoimmune disease
  * Ongoing infection (e.g., HIV or hepatitis)

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Prior radiation where the indicator lesion(s) are in the irradiated field
* Prior organ transplantation
* Participation in another clinical trial within 30 days prior to study entry
* Concurrent anticancer drugs/treatments or experimental medications
* Other concurrent investigational therapy
* Other concurrent chemotherapy, immunotherapy, or radiotherapy (including palliative radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy and tolerability of everolimus | Until treatment ends

SECONDARY OUTCOMES:
Evaluation of the efficacy of everolimus to induce molecular remission in patients treated with this regimen. | Until treament ends
Investigation of immunoglobulin heavy chain variable gene somatic hypermutations | Until treatment ends
  Investigation of immunoglobulin heavy chain variable gene somatic hypermutations (Ig-V_H) in classical mantle cell lymphoma as compared to blastoid mantle cell lymphoma, in particular in regard to their frequency, mutation distribution pattern (antigen selected vs. at random), and the individually involved Ig-V_H families.
Evaluation of a putative impact of Ig-V_H on clinical outcome. | Until treatment ends

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Renner, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (21):
- France (4):
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - University of Bologna Medical School, Bologna
  - European Institute of Oncology, Milan
- Switzerland (15):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopitaux Universitaires de Geneve, Thonex-Geneve
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum - Klinik im Park, Zurich
  - Klinik Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Renner C, Zinzani PL, Gressin R, Klingbiel D, Dietrich PY, Hitz F, Bargetzi M, Mingrone W, Martinelli G, Trojan A, Bouabdallah K, Lohri A, Gyan E, Biaggi C, Cogliatti S, Bertoni F, Ghielmini M, Brauchli P, Ketterer N; Swiss SAKK and French GOELAMS group from European Mantle Cell Lymphoma Network. A multicenter phase II trial (SAKK 36/06) of single-agent everolimus (RAD001) in patients with relapsed or refractory mantle cell lymphoma. Haematologica. 2012 Jul;97(7):1085-91. doi: 10.3324/haematol.2011.053173. Epub 2012 Feb 7. PMID 22315486